CLINICAL TRIAL: NCT06666738
Title: Evidence Based QUality Improvement for Prescribing Stewardship in ICU: Can a Structured Antimicrobial Review be Implemented in LMIC ICUs?
Brief Title: Evidence Based QUality Improvement for Prescribing Stewardship in ICU (EQUIPS-ICU)
Acronym: EQUIPS-ICU
Status: Not yet recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Nat Intensive Care Surveillence-MORU (Unknown)
Responsible Party: Sponsor
Other Study IDs: HCR24005 (559-24)
Record Dates: First submitted 2024-10-23; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Antimicrobial Stewardship
Keywords: Critical care; Antimicrobial Stewardship; Implementation; Quality improvement; Low or Middle Income Country (LMIC)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Structured antimicrobial review — The appropriateness of the documented indication, route of administration, expected duration and stop date of all antimicrobials will be reviewed within 48 hours of their prescription.

SUMMARY:
The goal of this observational study is to learn about the implementation of a process to review antimicrobial prescriptions for adult patients in Intensive Care Unit (ICU).

The main question it aims to answer is: can a structured antimicrobial review can be implemented in ICUs?

Implementation will be supported by the use of local protocols, audit and feedback, and education. It will be evaluated by daily data collection of clinical processes and interviews with local champions.

Resources to conduct the study are provided by the Wellcome Flagship Innovations award. ("Collaboration for Research, Implementation and Training in Critical Care in Asia and Africa", reference 224048/Z/21/Z).

ELIGIBILITY:
Inclusion Criteria:

* All adult ICUs within CCAA-affiliated Care Quality Registries
* ICUs must appoint a named Champion to facilitate implementation
* All antimicrobial prescriptions for adult patients within the ICUs described above

Exclusion Criteria:

• ICU's which demonstrate adoption and reach of 80% or greater (median over 2 months) of a pre-existing structured antimicrobial review

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All adult ICUs within CCAA-affiliated CQRs, where surveillance of antimicrobial utilisation has already been established will be considered for participation.
  ICUs must appoint a named Champion in order to participate. A survey will be conducted to determine pre-existing prescribing practice and the presence, characteristics and current adoption of structured review activities. Pre-existing antimicrobial review processes are neither a requirement for an ICU to participate nor an exclusion criterion. Instead, parallel to the survey, pre-implementation patient-level data pertaining to current antimicrobial prescribing review practices will be measured during months 1-2. ICU's which are found to already have a structured antimicrobial review in place, and which demonstrate adoption and reach of 80% or greater (median over the 2 months) will not be eligible to participate in the implementation to reduce confounding of the selected measures for implementation success.
Sampling Method: Non-Probability Sample
Enrollment: 6300 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Fidelity | Evaluated over calendar month periods during months 4-6 (i.e. the three months immediately following implementation)
  The proportion of prescriptions reviewed as intended (reviewed within 48hours with documentation of all 4 review components: indication, route, duration, stop date). Reported as a proportion of the number of possible reviews.
Reach | Evaluated over calendar month periods during months 4-6 (i.e. the three months immediately following implementation)
  Proportion of eligible patients who receive a review
Adoption | Evaluated over the calendar month period of month 7
  Proportion of prescriptions reviewed as intended once implementation support has been withdrawn

SECONDARY OUTCOMES:
Antimicrobial Density (AD) | Evaluated over calendar month periods during months 1-7 of the study.
  Defined Daily Dose / 1000 patient-days. This measure of antimicrobial consumption will compare prescribed daily doses of antimicrobials to those specified by the World Health Organization (WHO) (Anatomical Therapeutic Classification (ATC) J01 Defined Daily Doses). To correct for ICU unit size the investigators will standardise by number of admitted patient-days during that month in that ICU.
Duration of Therapy | Evaluated over calendar month periods during months 1-7 of the study
  Number of Days of antimicrobial Therapy / 1000 patient-days Analysed at the ICU level
Antimicrobial Redundancy Rate | Evaluated over calendar month periods during months 1-7 of the study
  Days of Therapy of prespecified redundant combinations of antimicrobials. Analysed at the ICU level.
Antimicrobial resistance rate | Evaluated over calendar month periods during months 1-7 of the study
  Number of multidrug-resistant pathogens (as specified by WHO priority list) / number of patients
Antimicrobial prescribing rate | Evaluated over calendar month periods during months 1-7 of the study
  Number of patients receiving at least 1 antimicrobial / number of patients admitted to ICU in the same period

CONTACTS AND LOCATIONS:
Overall Officials: Abi Beane, Dr., Principal Investigator — University of Oxford

IPD SHARING:
Plan to Share IPD: Yes
With participants' consent, as per the record of verbal consent, de-identified data may be uploaded to data repositories or shared with other researchers in line with MORU's data sharing policy.
Time Frame: After completion of the study
Access Criteria: Mahidol Oxford Tropical Medicine Research Unit (MORU) Data Sharing Policy
URL: https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing

REFERENCES:
- [Derived] Wagstaff D, Amuasi J, Arfin S, Aryal D, Nor MBM, Bonney J, Dondorp A, Dongelmans D, Dullawe L, Fazla F, Ghose A, Hanciles E, Haniffa R, Hashmi M, Smith AH, Kumar B, Minh YL, Moonesinghe R, Pisani L, Sendagire C, Hasan MS, Ghalib MS, Frimpong MS, Ranzani O, Sultan M, Thomson D, Tripathy S, Thwaites L, Uddin RAME, Mazlan MZ, Waweru-Siika W, Beane A. Evidence based QUality Improvement for Prescribing Stewardship in ICU (EQUIPS-ICU): protocol for type III hybrid implementation-effectiveness study. Implement Sci. 2025 Feb 25;20(1):12. doi: 10.1186/s13012-024-01413-4. PMID 40001051